CLINICAL TRIAL: NCT01173952
Title: Prospective Evaluation of Quality of Life in Men Undergoing Robotic Assisted Laparoscopic Radical Prostatectomy Vs. Radical Retropubic Prostatectomy
Brief Title: Quality of Life in Men Undergoing Robotic Assisted Laparoscopic Radical Prostatectomy Versus Radical Retropubic Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sung Won Lee, M.D.& Ph.D./Professor, Samsung Medical Center, Sungkyunkwan University School of Medicine, Department of Urology Samsung Medical Center, Sungkyunkwan University School of Medicine
Other Study IDs: 2010-06-026
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-06

CONDITIONS: Prostatic Neoplasms; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is prospective evaluation of quality of life in men undergoing robotic assisted laparoscopic radical prostatectomy versus radical retropubic prostatectomy.

DETAILED DESCRIPTION:
Preoperatively, enrolled patients will complete questionnaires called EPIC that will ask about urinary, sexual, bowel and hormonal function

At 1, 3,6,9 and 12 months after surgery, pateints will complete the questionnaires again.

All will be enrolled at Samsung Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of prostate adenocarcinoma
* Clinical stage: AJCC (VI) stage T1-T2 N0M0
* Primary treatment at Samsung Medical Center for prostate cancer using: radical retropubic prostatectomy, robotic prostatectomy

Exclusion Criteria:

* Clinical Stage: T3, T4, nodal or distant metastasis
* All kind of neoadjuvant, concurrent and adjuvant treatment
* poor health forced a patient into dropout

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Lee, M.D.& Ph.D., Study Chair — Department of Urology Samsung Medical Center